CLINICAL TRIAL: NCT03397888
Title: The Effect o f Hepatic Impairment on the Pharmacokinetics and Pharmacodynamics of Betrixiban, an Oral FXa Antagonist
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-022
Record Dates: First submitted 2017-12-07; First posted 2018-01-12 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Mild Impairment, Child-Pugh Category A
  Interventions: Drug: Betrixaban
- Cohort 2 (Experimental): Moderate Impairment, Child-Pugh Category B
  Interventions: Drug: Betrixaban
- Cohort 3 (Experimental): Essentially Healthy man or woman without liver disease matched to Cohorts 1 & 2 for age, sex and weight.
  Interventions: Drug: Betrixaban

INTERVENTIONS:
Drug: Betrixaban — 80 mg capsule

SUMMARY:
Single center, prospective open label PK and PD study of betrixaban in subjects with mild and moderate hepatic impairment vs healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Cohorts 1 & 2: Man or a woman 18 to 70 with stable chronic hepatic impairment disease due to cirrhosis confirmed by biopsy, ultrasound, CT or MRI (Cohort 1 - Mild impairment, Child-Pugh Category A; Cohort 2 - Moderate Impairment, Child-Pugh Category B). Cohort 3: essentially healthy man or woman without liver disease whose sex, age and weight match patients in Cohorts 1 & 2 in order to result in similar average demographics.
2. Body Mass Index between 18 and 35 kg*m-2 and weighs at least 50 kg.
3. Contraception. Men must agree to acceptable methods of contraception. Women of child-bearing potential must agree to two acceptable forms of contraception. Post-menopausal women must have had no regular menstrual bleeding for at least one year prior to initial dosing and confirmed by an elevated plasma Follicle-stimulating hormone level test at screening for women not in receipt of hormone replacement therapy (HRT). Women who report surgical sterilization must have had the procedure at least six months prior to dosing, supported by clinical documentation.
4. The subject has clinical unremarkable medical history, physical examination, ECG, laboratory values and vital signs, as determined by the investigator. Subjects in Cohorts 1 & 2 may have: abnormal liver function tests, INR up to 2.2, PT up to 6 seconds over control, aPPT up to 45 seconds and platelets down to 45,000/uL.
5. The subject smokes <12 cigarettes per day or equivalent and agrees to no or reduced tobacco products while domiciled.
6. The subject is able to read and give written informed consent and signed the IRB approved consent form.
7. The subject has adequate venous access for blood sampling.

Exclusion Criteria:

1. The subject has a history, symptoms of, or risk factors for bleeding or a stool specimen within 6 months of dosing positive for occult blood.
2. The subject has an absolute/relative contraindication to anticoagulation due to: history of intracranial bleeding, severe active bleeding, recent brain, eye, or spinal cord surgery or major surgery within 6 months of dosing.
3. The subject has a history of or risk factors for a hypercoagulable or thrombotic condition.
4. The subject has a history of any clinically significant cardiac, endocrinologic, hematologic, hepatic (except for Cohorts 1 & 2), immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal or other major disease other than the underlying disease in Cohorts 1 & 2.
5. The subject has a calculated creatinine clearance of <60mL/min as determined by Cockcroft-Gault method.
6. Concomitant medication use:

   1. For all subjects, illicit drugs, oral contraceptives, and hormone replacement therapy are excluded within 30 days prior to Day -1.
   2. For all subjects, over the counter drugs, including dietary supplements and herbal products are excluded within 14 days prior to Day -1.
   3. Subjects enrolled in Cohort 3 will be excluded if the subject has taken any prescription drugs in the 30 days prior to dosing. Furthermore, the subject will be excluded if he/she does not agree to refrain from concomitant drugs throughout the study unless medically necessary as determined by the Investigator.
   4. Subjects enrolled in Cohort 1 and 2 may continue taking stable preexisting medications throughout the study with the exception of strong P-gp inhibitors. Strong P-gp inhibitors include but are not limited to: amiodarone, azithromycin, clarithromycin, erythromycin, ketoconazole, and verapamil. Prescribed stable acetaminophen use up to 2,000 mg per day is allowable. Any acetaminophen use with alcohol within 48 hours of dosing is prohibited. Furthermore, the subject will be excluded if he/she does not agree to refrain from additional concomitant drugs throughout the study unless medically necessary as determined by the Investigator.
7. The subject has a history of severe trauma or bone fracture within 6 months prior to dosing; or planned surgery within 1 month after dosing.
8. The subject has a history of blood donation of more than 500mL within 3 months prior to dosing.
9. The subject has received an investigational drug product within 30 days or 5 half-lives of the investigational compound, whichever is greater, from Day -1.
10. The subject has positive screen for drugs of abuse at Day -1.
11. The subject does not agree to withhold from alcohol consumption from 48 hours prior to dosing through discharge.
12. The subject has a medical or surgical condition which may impair drug absorption.
13. The subject is pregnant or breastfeeding.
14. The subject has any condition which could interfere with or for which the treatment might interfere with the conduct of the study, or would, in the opinion of the Investigator, increase the risk of the subject's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
PK - Plasma half-life (t1/2) | Day 1 through Day 6
  Plasma half-life (t1/2), distribution half-life and terminal half-life.
PK - Tmax | Day 1 through Day 6
  Time to maximum observed plasma concentration (Tmax).
PK - Cmax | Day 1 through Day 6
  Maximum observed plasma concentration (Cmax)
PK - AUC (0-last) | Day 1 through Day 6
  Area under the plasma concentration-time curve from 0 to last measurable concentration (AUC (0-last)).
PK - (AUC(0-∞)). | Day 1 through Day 6
  Total area under the plasma concentration-time curve from time 0 to infinity (AUC(0-∞)).
PK - Volume of distribution | Day 1 through Day 6
  Apparent volume of distribution (Vd/F).
PK - Total clearance | Day 1 through Day 6
  Apparent total clearance (CL/F).

SECONDARY OUTCOMES:
Safety - Treatment Emergent AEs | Day -1 through up to Day 21
  Safety evaluation will study the adverse event (AE) profile
Safety - Demographics | Day -30 through Day -2 (Screening)
  Safety will be evaluated by assessment of Demographics
Safety - Vital Signs Temperature | Day -30 through up to Day 21
  Safety will be evaluated by assessment of Temperature - Celsius
Safety - Vital Signs Respiratory Rate | Day -30 through up to Day 21
  Safety will be evaluated by assessment of Respiratory Rate - Breaths per Minute
Safety - Vital Signs Heart Rate | Day -30 through up to Day 21
  Safety will be evaluated by assessment of Heart Rate - Beats per Minute
Safety - Vital Signs Blood Pressure | Day -30 through up to Day 21
  Safety will be evaluated by assessment of Blood Pressure - mmHg
Safety - 12 Lead ECG - PR | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - PR (ms)
Safety - 12 Lead ECG - RR | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - RR (ms)
Safety - 12 Lead ECG - WRS | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - WRS (ms)
Safety - 12 Lead ECG - QT | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - QT (ms)
Safety - 12 Lead ECG - QTcF | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - QTcF (ms)
Safety - 12 Lead ECG - QTcB | Day -30 through up to Day 21
  Safety will be evaluated by assessment of 12 ECG - QTcB (ms)
Safety - Physical Exam - Height | Day -30 through up to Day 21
  Safety will be evaluated by assessment Physical Exam - Height (centimeters)
Safety - Physical Exam - Weight | Day -30 through up to Day 21
  Safety will be evaluated by assessment Physical Exam - Weight (kilogram)
Safety - Lab - Hematology - hemoglobin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Hematology - hemoglobin (g/dL)
Safety - Lab - Hematology - hematocrit | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Hematology - hematocrit (%)
Safety - Lab - Hematology - white blood cell [WBC] | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Hematology - WBC (K/UL)
Safety - Lab - Hematology - Platelet Count | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Platelet Count (Plt/mL)
Safety - Lab - Hematology - Absolute Neutrophil Count | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Absolute Neutrophil Count (K/UL)
Safety - Lab - Hematology - Absolute Basophils | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Absolute Basophils (K/UL)
Safety - Lab - Hematology - Eosinophil's | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Eosinophil's (K/UL)
Safety - Lab - Hematology - Lymphocytes | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Lymphocytes (K/UL)
Safety - Lab - Hematology - Mean Corpuscular Hemoglobin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Mean Corpuscular Hemoglobin (PG)
Safety - Lab - Hematology - Mean Corpuscular Hemoglobin Concentration | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Mean Corpuscular Hemoglobin Concentration (g/dL)
Safety - Lab - Hematology - Mean Corpuscular Hemoglobin Volume | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Mean Corpuscular Hemoglobin Volume (FL)
Safety - Lab - Hematology - Monocytes | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Monocytes (K/UL)
Safety - Lab - Hematology - Neutrophils | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Neutrophils (K/UL)
Safety - Lab - Hematology - Red Blood Cell Count | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Red Blood Cell Count (MIL/UL)
Safety - Lab - Hematology - Red Cell Distribution Width | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Red Cell Distribution Width (%)
Safety - Lab - Hematology - Reticulocyte | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Reticulocyte (K/UL)
Safety- Lab - Coagulation - PT | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Coagulation - PT (seconds)
Safety- Lab - Coagulation - INR | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Coagulation - INR (no unit)
Safety- Lab - Coagulation - aPTT | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Coagulation - aPTT (seconds)
Safety- Lab - Coagulation - Factor V Leiden | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Coagulation - Factor V Leiden (positive/negative)
Safety - Lab - Serum Chemistry - Sodium | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Sodium (mEq/L)
Safety - Lab - Serum Chemistry - Potassium | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Potassium (mEq/L)
Safety - Lab - Serum Chemistry - Chloride | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Chloride (mEq/L)
Safety - Lab - Serum Chemistry - Carbon Dioxide | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Carbon Dioxide (mEq/L)
Safety - Lab - Serum Chemistry - Glucose | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Glucose (mg/dL)
Safety - Lab - Serum Chemistry - Blood Urea Nitrogen | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Blood Urea Nitrogen (mg/dL)
Safety - Lab - Serum Chemistry - Creatinine | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Creatinine (mg/dL)
Safety - Lab - Serum Chemistry - AST | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - AST (U/L)
Safety - Lab - Serum Chemistry - ALT | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - ALT (U/L)
Safety - Lab - Serum Chemistry - GGT | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - GGT (U/L)
Safety - Lab - Serum Chemistry - Total Protein | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Total Protein (g/dL)
Safety - Lab - Serum Chemistry - Albumin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Albumin(g/dL)
Safety - Lab - Serum Chemistry - Alkaline Phosphatase | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Alkaline Phosphatase (U/L)
Safety - Lab - Serum Chemistry - Calcium | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Calcium (mg/dL)
Safety - Lab - Serum Chemistry - Phosphorus | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Phosphorus (mg/dL)
Safety - Lab - Serum Chemistry - Total Bilirubin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Total Bilirubin (mg/dL)
Safety - Lab - Serum Chemistry - Fractionated Bilirubin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Fractionated Bilirubin(mg/dL)
Safety - Lab - Serum Chemistry - Uric Acid | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry - Uric Acid (mg/dL)
Safety - Lab - Serum Chemistry - LDH | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Chemistry LDH (U/L)
Safety - Lab - Urine toxicology Panel - Amphetamines | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Amphetamines (NG/ML)
Safety - Lab - Urine toxicology Panel - Barbiturates | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Barbiturates (NG/ML)
Safety - Lab - Urine toxicology Panel - Cannabinoids | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Cannabinoids (NG/ML)
Safety - Lab - Urine toxicology Panel - Cocaine | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Cocaine (NG/ML)
Safety - Lab - Urine toxicology Panel - Ethanol | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Ethanol (MG/DL)
Safety - Lab - Urine toxicology Panel - Opiates | Day -30 through Day -1
  Safety will be evaluated by analyzing Urine toxicology Panel - Opiates (NG/ML)
Safety - Lab - Urinalysis - Specific Gravity | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Specific Gravity (no unit)
Safety - Lab - Urinalysis - pH | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - pH (no unit)
Safety - Lab - Urinalysis - Glucose | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Glucose (no unit)
Safety - Lab - Urinalysis - Protein | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Protein (no unit)
Safety - Lab - Urinalysis - Hemoglobin | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Hemoglobin (no unit)
Safety - Lab - Urinalysis - Leukocyte esterase | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Leukocyte esterase (no unit)
Safety - Lab - Urinalysis - Nitrate | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Urinalysis - Nitrate (no unit)
Safety - Urine Occult Blood Testing | Day -30 through Day -2 (screening)
  Safety will be evaluated by assessment of Urine Occult Blood Testing (positive/negative)
Safety - Fecal Occult Blood Testing | Day -30 through Day -2 (screening)
  Safety will be evaluated by assessment of Fecal Occult Blood Testing (positive/negative)
Safety - Lab - Blood Virology - HIV I | Day-30 through Day -2 (Screening)
  Safety will be evaluated by analyzing Blood Virology - HIV I (positive/negative)
Safety - Lab - Blood Virology - HIV II | Day-30 through Day -2 (Screening)
  Safety will be evaluated by analyzing Blood Virology - HIV II (positive/negative)
Safety - Lab - Blood Virology - Hepatitis B | Day-30 through Day -2 (Screening)
  Safety will be evaluated by analyzing Blood Virology - Hepatitis B (positive/negative)
Safety - Lab - Blood Virology - Hepatitis C | Day-30 through Day -2 (Screening)
  Safety will be evaluated by analyzing Blood Virology - Hepatitis C (positive/negative)
Safety - Lab - Serum Pregnancy | Day -30 through up to Day 21
  Safety will be evaluated by analyzing Serum Pregnancy
PD - Anti-Factor Xa Concentration | Day 1 through Day 6
  Anti-fXa will be analyzed for changes/percent changes from baseline over time.
PD - Thrombin Concentrations | Day 1 through Day 6
  Thrombin will be analyzed for changes/percent changes from baseline over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States